CLINICAL TRIAL: NCT02824393
Title: Experimental Autologous Mesenchymal Stem Cell Therapy in Treatment of Chronic Autoimmune Urticaria
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Celal Bayar University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Acıbadem Labcell (Other)
Responsible Party: Principal Investigator, Cengiz Kırmaz, Professor Doctor (MD), Celal Bayar University
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: TUBITAK-1001-215S612
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Urticaria; Autoimmune Diseases; Immune System Diseases; Skin Diseases
Keywords: Mesenchymal stem cell; Chronic autoimmune urticaria
MeSH Terms: conditions — Urticaria; Autoimmune Diseases; Immune System Diseases; Skin Diseases; Chronic Urticaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal stem cell (Experimental): Intravenous infusion of ex vivo cultured adipose tissue derived autologous mesenchymal stem cells, twice at two week intervals in total 1x10/6 cells/kg.
  Interventions: Biological: Autologous mesenchymal stem cell
- Control patients (No Intervention): The patients who treated with the conventional therapy for urticaria, but not treat with mesenchymal stem cell.

INTERVENTIONS:
Biological: Autologous mesenchymal stem cell — Intravenous infusion of ex vivo cultured adipose tissue derived autologous mesenchymal stem cells, twice at two week intervals in total 1x10/6 cells/kg.
  Other Names: Autologous adipose tissue derived mesenchymal stem cell
  Arms: Mesenchymal stem cell

SUMMARY:
The aim of this study is to determine whether autologous adipose tissue derived Mesenchymal Stem Cells of treatment for chronic autoimmune urticaria is safe and effective.

DETAILED DESCRIPTION:
Chronic urticaria is a distressful disease, which negatively affects the quality of life. Pathogenesis isn't exactly clear, treatment is relatively palliative and results are usually suboptimal. 30-40% of the patients have autoimmune origin. Patients are forced to use immunosuppressive treatments which have systemic effects. Some of the treatments have effects as severe as the disease itself.

Mesenchymal stem cells (MSCs) are the most common used cells in clinical trials. These cells can provide efficient immunosuppression in severe conditions like immunosuppressive resistant Graft versus Host Disease. With this study at the first time and quite a different approach from conventional treatment, it will be tried an experimental treatment that used in the MSCs for the chronic autoimmune urticaria patients without of definitive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with chronic autoimmune urticaria (at least six months before)
2. Patients who have >20 and over of urticaria activity score [according to European Academy of Allergy and Clinical Immunology (EAACI) / Global Allergy and Asthma European Network (GALEN) guidelines].
3. Patients who capable of own daily findings record.
4. Patients who could not be controlled despite the use of a treatment agent in the fourth step for 3 months (according to EAACI / GALEN guidelines).

Exclusion Criteria:

1. Patients who have heart, liver or renal failure.
2. Patients who have epilepsy, cerebrovascular or ischemic attack.
3. Patients who have atopic dermatitis or another underlying itchy skin disease.
4. Patients who have parasitic infection.
5. Patients who have antibiotic allergy.
6. History of malignancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly urticaria activity scores. | 6 months
  The weekly urticaria activity scores will be assessed according to European Academy of Allergy and Clinical Immunology (EAACI) / Global Allergy and Asthma European Network (GALEN) guidelines.

SECONDARY OUTCOMES:
Follow-up of the mesenchymal stem cell treatment-related side effects according to World Health Organisation (WHO) Toxicity Grading Scale for Determining The Severity of Adverse Events. | 12 months
The changes in the ratios of peripheral blood cluster of differentiation 4 (CD4) T cell subsets. | 6 months
The changes in ratios of peripheral blood inflammatory and anti-inflammatory cytokines. | 6 months
The changes in the levels of peripheral blood anti-FcεRI autoantibody | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alper Tunga Özdemir, PhD, Principal Investigator — Ege University, Institute of Health Sciences, Department of Stem Cell, Izmir/TURKEY; Ercüment Ovalı, Prof. Dr., Principal Investigator — Acıbadem Labcell, Istanbul/TURKEY
Locations (1):
- Celal Bayar University, Medical School, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes